CLINICAL TRIAL: NCT00172510
Title: Mutation Analysis of 17α-Hydroxylase
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701060
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-08

CONDITIONS: Pseudohermaphroditism; Congenital Adrenal Hyperplasia; Hypertension
MeSH Terms: conditions — Disorders of Sex Development; Adrenal Hyperplasia, Congenital; Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: blood drawing

SUMMARY:
To elucidate the molecular pathology of the 4 families with 17α-hydroxylase/17,20-lyase deficiency.

DETAILED DESCRIPTION:
17α-hydroxylase is a rare form of congenital adrenal hyperplasia. Patients with complete 17α-hydroxylase deficiency may come to attention to the doctor at their early adulthood due to hypertension or disordered puberty. 17α-hydroxylase is a form of cytochrome P450 enzyme in the adrenal cortex for the production of cortisol, while 17,20-lyase is required in both adrenal glands and the gonads for the production of androgen precursors of sex hormones. Therefore, patients with 17α-hydroxylase will presented with elevated deoxycorticosterone (DOC) level and decreased aldosterone and cortisol level. Because DOC is the second most important naturally occurring mineralocorticoid hormone, hypertension and hypokalemic alkalosis will be noted in these patients. Besides, deficiency of 17,20-lyase activity will lead to impairment of virilization in 46 XY patients and deficient estrogen production in 46 XX patients.

The P450c17 has both 17α-hydroxylase and 17,20-lyase activity and are encoded by the CYP17 gene. The sequence of CYP17 gene was established in 1987 and more than 40 mutations were identified till now. The purpose of this study is to elucidate the molecular pathology of the 4 families with 17α-hydroxylase/17,20-lyase deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 17α-hydroxylase deficiency and their family

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2004-08; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ching Tung, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan